CLINICAL TRIAL: NCT01287962
Title: Apatinib in the Treatment of Advanced Non-squamous Non-small Cell Lung Cancer:a Randomised, Double-blind, Placebo-controlled, Multicentre Phase III Study
Brief Title: Apatinib in the Treatment of Advanced Non-squamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HENGRUI 20110301
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2012-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Apatinib; Non-small Cell Lung Cancer; VEGFR TKIs
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apatinib (Experimental): 750 mg，po，QD； 28 days every cycle
  Interventions: Drug: apatinib
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: apatinib — 750 mg，po，QD； 28 days every cycle
  Arms: Apatinib
Drug: placebo — po，QD； 28 days every cycle
  Arms: Placebo

SUMMARY:
Apatinib is a new kind of Vascular endothelial growth factor receptor(VEGFR) tyrosine kinase inhibitors (TKIs). The investigators have finished the preclinical and phase I and phase II clinical study for apatinib and found its satisfactory anti-tumor activity and tolerated toxicities. A disease-control rate of 75% was found in lung cancer patients. In the present phase III trial, the investigators will further evaluate the efficacy and toxicities of apatinib in the treatment of advanced non-squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 to 70 years of age
2. Documented pathological evidence of advanced non-squamous non-small cell lung cancer with measurable lesions
3. Failure of epidermal-growth-factor receptor (EGFR) TKIs target treatment and second-line or more regimens of chemotherapy
4. Eastern Cooperative Oncology Group (ECOG) performance status between 0 and 1
5. Patients had to have recovered from any toxic effects of therapy
6. Patients with brain/meninges metastasis should keep stable disease for 2 months before randomisation
7. Adequate hematologic and biochemical values were required

Exclusion Criteria:

1. Presence of small-cell lung cancer alone or with NSCLC
2. Pregnant or breast-feeding women
3. Severe or uncontrolled systemic disease such as clinically significant hypertension(systolic pressure > 140 mmHg，diastolic pressure > 90 mmHg), cardiac ischemia and infarction, ventricular arrhythmias(QT ≥ 440ms) and grade 1 cardiac insufficiency
4. Difficulties in taking pills (inability to swallow tablets,GI tract resection, chronic bacillary diarrhea and intestinal obstruction)
5. Coagulation disfunction,hemorrhagic tendency or receiving anticoagulant therapy
6. ≥ CTCAE 2 pneumorrhagia or ≥ CTCAE 3 hemorrhage in other organs within 4 weeks
7. Bone fracture or wounds that was not cured for a long time
8. Arterial thrombus or phlebothrombosis within 6 months and taking anticoagulant agents
9. Mental diseases and psychotropic substances abuse
10. Previous treatment with an experimental agent within 4 weeks
11. Previous treatment with VEGFR、platelet derived growth factor receptor(PDGFR) TKIS
12. Other coexisting malignant disease (apart from basal-cell carcinoma and carcinoma in situ of uterine cervix)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 24 months
  Progression-free survival as the time from randomization to documented disease progression according to response evaluation criteria in solid tumors (RECIST) or death.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 24 months
  ORR was the percentage of patients who got partial or complete response
Overall Survival(OS) | 24 months
  OS was determined from date of enrollment until death or the date the patient was recorded alive of last follow-up
Toxicity | 24 months
  Adverse events (AEs) were recorded, graded for toxicity using the NCI-CTC, and assessed by the investigator for any relationship with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Study Chair — Cancer Center of Sun Yat-Sen University (CCSU)
Locations (1):
- Cancer Center of Sun Yat-Sen University (CCSU), Guangzhou, Guangdong, China